CLINICAL TRIAL: NCT02645968
Title: Registry for Exploring Clinical and Epidemiological Characteristics of Interstitial Lung Diseases - EXCITING
Acronym: EXCITING
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Collaborators: University of Giessen (Other); German Center for Lung Research (Other); Helmholtz Zentrum München (Industry); Institut für Lungenforschung e.V. (Unknown); German Respiratory Society (Other); WATL e.V. (Unknown); Bundesverband der Pneumologen (Unknown); Lungenfibrose e.V. (Unknown); Sacura GmbH (Other); Syneed Medidata GmbH (Industry)
Responsible Party: Principal Investigator, Michael Kreuter, Head of Center for interstitial and rare lung diseases, Heidelberg University
Other Study IDs: ILD Patient Registry
Record Dates: First submitted 2015-12-28; First posted 2016-01-05 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Interstitial Lung Disease (ILD)
Keywords: Pneumology; Registry; EXCITING; Interstitial lung disease; ILD
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect valid data from all forms of health care on the incidence, prevalence, the regional distribution, characteristics, management and outcomes of different ILDs under clinical practice conditions.

DETAILED DESCRIPTION:
Interstitial lung diseases (ILD) are a heterogeneous group of more than 200 entities that can be idiopathic or as a result of other diseases and/or treatments. All forms of ILD are considered to be seldom or very seldom (and most of them are so-called "orphan" diseases), in their entirety they seem to represent an epidemiological burden, which should not be underestimated, e.g. as "normal" symptoms of the elderly.

The knowledge about the epidemiology of ILDs is very limited, in general and in Germany in particular. For Germany no current, valid and comprehensive population-based data on ILDs exist because no appropriate ILD classification was available for a long time. The epidemiological data, which were collected before the introduction of the current classification of ILD according to the ATS/ERS consensus and before HRCT was considered the diagnostic gold standard, are not very reliable. Furthermore systemic investigations relating to the development of an ILD of risk groups, such as patients undergoing radio- or chemotherapy or patients with connective tissue disease, are restricted.

Thus, only little is known about costs associated with ILDs. Idiopathic Pulmonary Fibrosis (IPF), as one of the disease entities, was shown to be associated with high healthcare utilization and costs in England and the USA, as in many cases lung transplantation is the only therapeutic option and also new pharmaceutical treatments are costly. But there is a lack of data on healthcare utilization and financial consequences of other ILD than IPF in Germany. Therefore, this registry will provide an important database for health economics and health services research questions.

Against this background, this multi-centre, non interventional prospective observational disease and outcomes registry for ILD aims to collect valid data from all forms of health care on the incidence, prevalence, the regional distribution, characteristics, management and outcomes of different ILDs under clinical practice conditions. In detail, demographic data such as gender, age, country of birth, place of residence; disease related data such as subtype of ILD, treatment center, diagnostic procedures (e.g. HRCT, lung biopsy, pulmonary function tests); risk factors (e.g. smoking status, profession, familial ILD); co-morbidities; ILD management as analysed by the kind and frequency of pharmacological and non-pharmacological therapies; outcome; and consumption of resources will be recorded. Therefore, this registry will allow obtaining a comprehensive and current epidemiologic report for ILDs in Germany and can be particularly helpful in uncovering correlations between risk exposure and disease development.

This study, with up to 100 sites, initially focused on the federal states Baden-Wuerttemberg and Hesse, is planned for a minimum of 5 years and 600 patients should be enrolled as part of the study a screening/baseline visit, on which the Informed Consent Form will be signed, and every 6 months regularly updates/phone contacts will be performed.

Following quality procedures are applicable for this registry:

* Quality assurance plan that addresses data validation and registry procedures, including any plans for site monitoring and auditing.
* Data checks to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.
* Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources (e.g., medical records, paper or electronic case report forms, or interactive voice response systems).
* Standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management.
* Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect.
* Plan for missing data to address situations where variables are reported as missing, unavailable, "non-reported," uninterpretable, or considered missing because of data inconsistency or out-of-range results
* Statistical analysis plan describing the analytical principles and statistical techniques to be employed in order to address the primary and secondary objectives, as specified in the study protocol or plan.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Able to read and understand the scope and nature of data collection
* Aged ≥ 18 at time of informed consent
* Patients diagnosed with interstitial lung disease (ILD). Patients with suspicion on interstitial lung disease cannot be included into the registry, only after consens diagnosis of an ILD. This is also the case for patients with not classifiable ILDs.

Subjects with the following subtypes of ILD will be enrolled:

1. Idiopathic interstitial pneumonia (IIPs)

   * Idiopathic pulmonary fibrosis (IPF)
   * Non-specific interstitial pneumonia (NSIP)
   * Desquamative interstitial pneumonia (DIP)
   * Respiratory bronchiolitis-associated interstitial lung disease (RB-ILD)
   * Cryptogenic organizing pneumonia (COP)
   * Lymphocytic interstitial pneumonia (LIP)
   * Acute interstitial pneumonia (AIP)
   * Rare forms of IIPs (e.g. pleuropulmonary fibroelastosis)
   * Not classifiable IIP
2. Granulomatous lung disease

   * Sarcoidosis
   * Berylliosis
   * Other (e.g. involvement in chronic inflammatory liver and gut diseases, except EAA)
3. Hypersensitivity pneumonitis (exogen allergic alveolitis (EAA))

   * Farmer's lung
   * Bird keepers' lung disease
   * Origin unknown
   * Other
4. Rheumatic and connective tissue diseases with pulmonary involvement like:

   * Connective tissue disease (subtype)
   * Vasculitis
   * Rheumatoid arthritis
5. Pneumoconiosis

   * Asbestosis
   * Silicosis
   * Other
6. Other forms

   * Pulmonary lymphangioleiomyomatosis
   * Pulmonary Langerhans' cell histiocytosis
   * Pulmonary alveolar proteinosis
   * Eosinophilic pneumonia
   * Post-ARDS Fibrosis
7. Drug-related
8. Radiotherapy associated
9. Fibrosis in emphysema patients without signs of other ILDs (i.e. smoking related interstitial fibrosis or "emphysemasclerosis")
10. Others
11. Not classifiable

Furthermore for each subtype it will be queried, if a diagnosis of concomitant emphysema in ILD was made.

Exclusion Criteria:

- Patients without interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ILD patients from all forms of health care
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2014-05; Primary Completion 2020-04 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Determination of characteristics, management and outcomes of patients with different ILDs under clinical practice conditions. | Six month interval over 5 years
  1. (disease-related) characteristics of ILD patients
  2. diagnostic procedures for the identification of ILDs
  3. the clinical management of different (sub) types of ILD under clinical practice
  4. the outcome of different types of ILDs and of ILD related therapies from all forms of health care facilities

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kreuter, Prof. Dr., Principal Investigator — Centre for interstitial and rare lung diseases, Pneumology and Respiratory Medicine, Thorax Clinic, University Hospital Heidelberg
Locations (22):
- Germany (22):
  - Lungenärztliche Gemeinschaftspraxis Dr. Storz / Dr. Prettner, Böblingen, Baden-Wurttemberg
  - Thoraxklinik Heidelberg, Abteilung Pneumologie und Beatmungsmedizin, Heidelberg, Baden-Wurttemberg
  - Gesundheitsverbund Landeskreis Konstanz, Krankenhausbetriebsgesellschaft Konstanz, Konstanz, Baden-Wurttemberg
  - Pneumologische Praxis im Zentrum - PiZ, Dr. med. Hans-Paul Eulenbruch und Dr. med. Alexander Rupp, Stuttgart, Baden-Wurttemberg
  - Klinikum Stuttgart, Klinik für Allgemeine Innere Medizin, Gastroenterologie, Hepatologie und Infektiologie, Pneumologie, Stuttgart, Baden-Wurttemberg
  - Lungenpraxis Tübingen, Tübingen, Baden-Wurttemberg
  - Pneumologisches Zentrum, Wiesloch, Baden-Wurttemberg
  - Klinikverbund Kempten-Oberallgäu, Klinik für Pneumologie, Thoraxonkologie, Schlaf- und Beatmungsmedizin, Immenstadt im Allgäu, Bavaria
  - Pneumologische Gemeinschaftspraxis Fulda Dres. Wiederhold, Schratz, Wissner, Fulda, Hesse
  - Klinikum Fulda gAG, Medizinische Klinik V - Pneumologie, Fulda, Hesse
  - Universitätsklinikum Gießen und Marburg GmbH, Medizinische Klinik und Poliklinik II, Giessen, Hesse
  - Lungenfachklinik Immenhausen, Immenhausen, Hesse
  - Universitätsklinikum Aachen, Medizinische Klinik I, Aachen, North Rhine-Westphalia
  - Medizinisches Versorgungszentrum Malteser Bonn gem. GmbH, Malteser Lungen- und Allergiezentrum Bonn, Bonn, North Rhine-Westphalia
  - St. Marien-Hospital GmbH, Cologne, North Rhine-Westphalia
  - Malteser Krankenhaus St. Hildegardis, Klinik für Pneumologie und Beatmungsmedizin, Cologne, North Rhine-Westphalia
  - Johanniter-Krankenhaus Rheinhausen GmbH, Duisburg, North Rhine-Westphalia
  - Ruhrlandklinik - Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen, North Rhine-Westphalia
  - Klinkum Gütersloh, Medizinische Klink III, Pneumologie, Schlaf- und Beatmungsmedizin, Infektiologie und Allgemeine Innere Medizin, Gütersloh, North Rhine-Westphalia
  - Katholische Kranken- und Pflegeeinrichtung Leverkusen GmbH, St. Remigius Krankenhaus Opladen, Leverkusen, North Rhine-Westphalia
  - framol-med GmbH, Pneumoglische Gemeinschaftspraxis Rheine, Rheine, North Rhine-Westphalia
  - Krankenhaus Bethanien gGmbH, Klinik für Pneumologie und Allergologie, Zentrum für Schlaf- und Beatmungsmedizin, Solingen, North Rhine-Westphalia

REFERENCES:
- [Background] Demedts M, Wells AU, Anto JM, Costabel U, Hubbard R, Cullinan P, Slabbynck H, Rizzato G, Poletti V, Verbeken EK, Thomeer MJ, Kokkarinen J, Dalphin JC, Taylor AN. Interstitial lung diseases: an epidemiological overview. Eur Respir J Suppl. 2001 Sep;32:2s-16s. PMID 11816822
- [Background] Akgun KM, Crothers K, Pisani M. Epidemiology and management of common pulmonary diseases in older persons. J Gerontol A Biol Sci Med Sci. 2012 Mar;67(3):276-91. doi: 10.1093/gerona/glr251. Epub 2012 Feb 15. PMID 22337938
- [Background] Ferreira JP, Almeida I, Marinho A, Cerveira C, Vasconcelos C. Anti-ro52 antibodies and interstitial lung disease in connective tissue diseases excluding scleroderma. ISRN Rheumatol. 2012;2012:415272. doi: 10.5402/2012/415272. Epub 2012 Mar 27. PMID 22567412
- [Background] Gunnarsson R, Aalokken TM, Molberg O, Lund MB, Mynarek GK, Lexberg AS, Time K, Dhainaut AS, Bertelsen LT, Palm O, Irgens K, Becker-Merok A, Nordeide JL, Johnsen V, Pedersen S, Proven A, Garabet LS, Gran JT. Prevalence and severity of interstitial lung disease in mixed connective tissue disease: a nationwide, cross-sectional study. Ann Rheum Dis. 2012 Dec;71(12):1966-72. doi: 10.1136/annrheumdis-2011-201253. Epub 2012 May 1. PMID 22550317
- [Background] Hallowell RW, Reed RM, Fraig M, Horton MR, Girgis RE. Severe pulmonary hypertension in idiopathic nonspecific interstitial pneumonia. Pulm Circ. 2012 Jan-Mar;2(1):101-6. doi: 10.4103/2045-8932.94842. PMID 22558525
- [Background] Kobayashi A, Okamoto H. Treatment of interstitial lung diseases associated with connective tissue diseases. Expert Rev Clin Pharmacol. 2012 Mar;5(2):219-27. doi: 10.1586/ecp.12.9. PMID 22390563
- [Background] Tzouvelekis A, Galanopoulos N, Bouros E, Kolios G, Zacharis G, Ntolios P, Koulelidis A, Oikonomou A, Bouros D. Effect and safety of mycophenolate mofetil or sodium in systemic sclerosis-associated interstitial lung disease: a meta-analysis. Pulm Med. 2012;2012:143637. doi: 10.1155/2012/143637. Epub 2012 May 10. PMID 22655194
- [Background] Amar RK, Jick SS, Rosenberg D, Maher TM, Meier CR. Drug-/radiation-induced interstitial lung disease in the United Kingdom general population: incidence, all-cause mortality and characteristics at diagnosis. Respirology. 2012 Jul;17(5):861-8. doi: 10.1111/j.1440-1843.2012.02187.x. PMID 22563933
- [Background] King TE Jr. Smoking and subclinical interstitial lung disease. N Engl J Med. 2011 Mar 10;364(10):968-70. doi: 10.1056/NEJMe1013966. No abstract available. PMID 21388315
- [Background] Lederer DJ, Enright PL, Kawut SM, Hoffman EA, Hunninghake G, van Beek EJ, Austin JH, Jiang R, Lovasi GS, Barr RG. Cigarette smoking is associated with subclinical parenchymal lung disease: the Multi-Ethnic Study of Atherosclerosis (MESA)-lung study. Am J Respir Crit Care Med. 2009 Sep 1;180(5):407-14. doi: 10.1164/rccm.200812-1966OC. Epub 2009 Jun 19. PMID 19542480
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Background] Doyle TJ, Hunninghake GM, Rosas IO. Subclinical interstitial lung disease: why you should care. Am J Respir Crit Care Med. 2012 Jun 1;185(11):1147-53. doi: 10.1164/rccm.201108-1420PP. Epub 2012 Feb 23. PMID 22366047
- [Background] Lynge E. Implication for epidemiology of disease registers. Public Health Rev. 1993-1994;21(3-4):263-70. PMID 8047653
- [Background] American Thoracic Society; European Respiratory Society. American Thoracic Society/European Respiratory Society International Multidisciplinary Consensus Classification of the Idiopathic Interstitial Pneumonias. This joint statement of the American Thoracic Society (ATS), and the European Respiratory Society (ERS) was adopted by the ATS board of directors, June 2001 and by the ERS Executive Committee, June 2001. Am J Respir Crit Care Med. 2002 Jan 15;165(2):277-304. doi: 10.1164/ajrccm.165.2.ats01. No abstract available. PMID 11790668
- [Background] Demedts M, Costabel U. ATS/ERS international multidisciplinary consensus classification of the idiopathic interstitial pneumonias. Eur Respir J. 2002 May;19(5):794-6. doi: 10.1183/09031936.02.00492002. No abstract available. PMID 12030715
- [Background] Kreuter M, Herth FJ, Wacker M, Leidl R, Hellmann A, Pfeifer M, Behr J, Witt S, Kauschka D, Mall M, Gunther A, Markart P. Exploring Clinical and Epidemiological Characteristics of Interstitial Lung Diseases: Rationale, Aims, and Design of a Nationwide Prospective Registry--The EXCITING-ILD Registry. Biomed Res Int. 2015;2015:123876. doi: 10.1155/2015/123876. Epub 2015 Nov 10. PMID 26640781